CLINICAL TRIAL: NCT06408857
Title: A Phase 1b, Age De-Escalation/Dose Escalation Trial to Evaluate Safety, Tolerability, and Pharmacokinetics of MAM01 in an African Population of Adults and Children in a Setting of Perennial Malaria Transmission
Brief Title: Study To Evaluate Safety, Tolerability, and Pharmacokinetics of MAM01 in African Population
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gates Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gates MRI-MAM01-103
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: Malaria; Plasmodium falciparum; MAM01; De-Escalation; Dose Escalation; Perennial Malaria Transmission; Antibody; Monoclonal; Prevention; Pediatric; mAb-1797
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A: Open Label. Part B: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part A: Cohort 1a (Healthy Adults): 300 milligrams (mg) MAM01 subcutaneously (SC) (Experimental): Participants will receive MAM01.
  Interventions: Drug: MAM01 300 mg SC
- Part A: Cohort 1b (Healthy Adults): 300 mg MAM01 intramuscularly (IM) (Experimental): Participants will receive MAM01.
  Interventions: Drug: MAM01 300 mg IM
- Part A: Cohort 1c (Healthy Adults): 2000 mg MAM01 intravenously (IV) (Experimental): Participants will receive MAM01.
  Interventions: Drug: MAM01 2000 mg IV
- Part B: Cohort 2a (Healthy Younger Children): 190 mg MAM01 or placebo SC (Experimental): Participants will be randomized in 3:1 ratio (MAM01 : PBO)
  Interventions: Drug: MAM01 190 mg SC; Drug: Placebo SC
- Part B: Cohort 2b (Healthy Younger Children): 225 mg MAM01 or placebo SC (Experimental): Participants will be randomized in 3:1 ratio (MAM01 : PBO)
  Interventions: Drug: MAM01 225 mg SC; Drug: Placebo SC
- Part B: Cohort 3a (Healthy Infants): 150 mg MAM01 or placebo SC (Experimental): Participants will be randomized in 3:1 ratio (MAM01 : PBO)
  Interventions: Drug: MAM01 150 mg SC; Drug: Placebo SC
- Part B: Cohort 3b (Healthy Infants): 150 mg MAM01 or placebo IM (Experimental): Participants will be randomized in 3:1 ratio (MAM01 : PBO)
  Interventions: Drug: MAM01 150 mg IM; Drug: Placebo IM
- Part B: Cohort 3c (Healthy Infants): 150 mg MAM01 or placebo IV (Experimental): Participants will be randomized in 3:1 ratio (MAM01 : PBO)
  Interventions: Drug: MAM01 150 mg IV; Drug: Placebo IV
- Part B: Cohort 4a (Healthy Infants): 150 mg MAM01 or placebo SC (Experimental): Participants will be randomized in 3:1 ratio (MAM01 : PBO)
  Interventions: Drug: MAM01 150 mg SC; Drug: Placebo SC
- Part B: Cohort 4b (Healthy Infants): 150 mg MAM01 or placebo IM (Experimental): Participants will be randomized in 3:1 ratio (MAM01 : PBO)
  Interventions: Drug: MAM01 150 mg IM; Drug: Placebo IM
- Part B: Cohort 4c (Healthy Infants): 150 mg MAM01 or placebo IV (Experimental): Participants will be randomized in 3:1 ratio (MAM01: PBO)
  Interventions: Drug: MAM01 150 mg IV; Drug: Placebo IV

INTERVENTIONS:
Drug: MAM01 300 mg SC — MAM01 300 mg will be administered SC
  Arms: Part A: Cohort 1a (Healthy Adults): 300 milligrams (mg) MAM01 subcutaneously (SC)
Drug: MAM01 300 mg IM — MAM01 300 mg will be administered IM route
  Arms: Part A: Cohort 1b (Healthy Adults): 300 mg MAM01 intramuscularly (IM)
Drug: MAM01 2000 mg IV — MAM01 2000 mg will be administered IV
  Arms: Part A: Cohort 1c (Healthy Adults): 2000 mg MAM01 intravenously (IV)
Drug: MAM01 190 mg SC — MAM01 190 mg will be administered SC
  Arms: Part B: Cohort 2a (Healthy Younger Children): 190 mg MAM01 or placebo SC
Drug: MAM01 225 mg SC — MAM01 225 mg will be administered SC
  Arms: Part B: Cohort 2b (Healthy Younger Children): 225 mg MAM01 or placebo SC
Drug: MAM01 150 mg SC — MAM01 150 mg will be administered SC
  Arms: Part B: Cohort 3a (Healthy Infants): 150 mg MAM01 or placebo SC; Part B: Cohort 4a (Healthy Infants): 150 mg MAM01 or placebo SC
Drug: MAM01 150 mg IM — MAM01 150 mg will be administered IM
  Arms: Part B: Cohort 3b (Healthy Infants): 150 mg MAM01 or placebo IM; Part B: Cohort 4b (Healthy Infants): 150 mg MAM01 or placebo IM
Drug: MAM01 150 mg IV — MAM01 150 mg will be administered IV
  Arms: Part B: Cohort 3c (Healthy Infants): 150 mg MAM01 or placebo IV; Part B: Cohort 4c (Healthy Infants): 150 mg MAM01 or placebo IV
Drug: Placebo SC — Placebo will be administered SC
  Arms: Part B: Cohort 2a (Healthy Younger Children): 190 mg MAM01 or placebo SC; Part B: Cohort 2b (Healthy Younger Children): 225 mg MAM01 or placebo SC; Part B: Cohort 3a (Healthy Infants): 150 mg MAM01 or placebo SC; Part B: Cohort 4a (Healthy Infants): 150 mg MAM01 or placebo SC
Drug: Placebo IV — Placebo will be administered IV.
  Arms: Part B: Cohort 3c (Healthy Infants): 150 mg MAM01 or placebo IV; Part B: Cohort 4c (Healthy Infants): 150 mg MAM01 or placebo IV
Drug: Placebo IM — Placebo will be administered IM
  Arms: Part B: Cohort 3b (Healthy Infants): 150 mg MAM01 or placebo IM; Part B: Cohort 4b (Healthy Infants): 150 mg MAM01 or placebo IM

SUMMARY:
This study will test a new drug (MAM01) to find which doses are safe and could help prevent people from getting malaria for at least 4 months. The study will take place in parts of Africa where malaria is common. Part A is an open-label study conducted in healthy adults whereas Part B is double-blind study conducted in young children and infants. Both the parts will evaluate the safety, tolerability and pharmacokinetics of MAM01.

DETAILED DESCRIPTION:
This is a Phase 1b, age de-escalation/dose escalation trial that will be conducted in a setting of perennial Plasmodium falciparum (malaria parasite) transmission in Africa. The study will be conducted in 2 parts: Part A (Dose Escalation in Adults); Part B (Age De-escalation/Dose Escalation in Younger Children and infants).

ELIGIBILITY:
Inclusion Criteria:

PART A

* Male or female adults aged 18 to 55 years inclusive at the time of signing the informed consent form (ICF), who are capable of, and willing to provide, informed consent
* Healthy, as determined by Investigator assessment, including medical history, physical examination, and screening laboratory results
* All dosing groups: hemoglobin level ≥ 8 grams per deciliter (g/dL)
* All dosing groups: living within local jurisdiction of trial site(s) and available for the duration of the trial for all cohorts
* Female participants of childbearing potential must be nonpregnant and agree to avoid becoming pregnant by using an acceptable contraception method

PART B

* Age Cohort 2: male or female children aged 2 years to <5 years at the time their parent or Legally Authorized Representative (LAR) signs the ICF
* Age Cohort 3: male or female children aged 12 months to <24 months at the time their parent or LAR signs the ICF
* Age Cohort 4: male or female infant children aged 3 months to <12 months and weighing at least 5 kilograms (kg) at the time their parent or LAR signs the ICF
* Healthy, as determined by Investigator assessment, including medical history, physical examination, and screening laboratory results
* Hemoglobin level ≥ 8g/dL
* Height and weight Z-scores ≥-2
* Living within local jurisdiction of trial site(s) and available for the duration of the trial

Exclusion Criteria:

PART A & PART B

* Within 48 hours prior to randomization, acute febrile illness

  * Sickle cell disease or history of splenectomy
  * Use of antimalarial chemoprevention or treatment, and/or antibiotics with known antimalarial effects (eg, clotrimoxazole, azithromycin, tetracyclines) within 30 days prior to dosing
  * Enrolled in another clinical trial within 90 days prior to Screening or planning to participate in another trial during, or within 1 year following, their participation in this trial
  * Received any doses of a malaria vaccine or other monoclonal antibodies (mAb) to Pf
  * Eligible to receive a malaria vaccine (RTS, S/AS01 or R21/Matrix-M) at screening or if it is expected to become available during the period of the trial.
  * History of allergy or hypersensitivity or contraindications to trial drugs (including those used as empirically treatment for Pf to clear any existing parasitemia), excipients or related substances
  * Any history of severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis prior to enrollment that has a reasonable risk of recurrence during the trial
  * History of any autoimmune disease or immunodeficiency or other impairment to the immune system, including HIV infection
  * Use of chronic (≥ 14 days) immunosuppressive agents including systemic steroids (eg, prednisone >10 milligrams per day [mg/day]) within 30 days prior to dosing. Use of inhaled or topical corticosteroids is permitted
  * Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising with blood draws
  * Receipt of immunoglobulins and/or blood products within the past 6 months
  * Any current uncontrolled medical or psychiatric condition, or substance abuse problems that in the opinion of the Investigator, will make it unlikely for participant to comply with the protocol, may interfere with study assessments, or could jeopardize the safety of the participant
  * Any contraindication for a subcutaneous injection, intravenous injection, or intramuscular injection, as applicable
  * For Part A, female participants who are breastfeeding, pregnant, or unable or unwilling to adhere to required contraception
  * For Part B, in the opinion of the Investigator, the parent or LAR may not be able to ensure participant compliance with the requirements of the trial

Ages: 3 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 123 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting Treatment-emergent adverse events (TEAEs) | Up to 28 days post dose (Part A and B)
Number of participants reporting serious adverse events (SAEs), adverse events of special interest (AESI), and AEs leading to discontinuation | Up to 182 days post dose
Number of participants reporting solicited systemic AEs and solicited injection site AEs (applicable to IM dosing) | Up to 7 days post dose
Number of participants reporting solicited systemic AEs and solicited injection site AEs (applicable to SC dosing) | Up to 7 days post dose

SECONDARY OUTCOMES:
Percentage of participants with graded abnormal clinical hematology and chemistry laboratory results | Up to 28 days post dose
Maximal observed blood concentration of MAM01 following the first dose (Cmax1) | Pre- and post-dose (IV dosing groups only) at Day 1, 4, 7, 14, 28, 56, 84, 112, 140, and 182
  Capillary blood samples will be collected for the analysis pharmacokinetic parameters. Blood concentrations of MAM01 will be measured using a validated immunoassay.
Concentration at Day 182 (C182) | At Day 182 post first dose
Total Area Under the Concentration Curve (AUC) Day 0 - Day 182 | From 0 to 182 days post dose
Percentage of participants with antidrug antibodies (ADAs) to MAM01 | At Days 1, 28, 84, and 182

CONTACTS AND LOCATIONS:
Locations (2):
- Uganda (2):
  - JCRC-Joint Clinical Research Centre, Kampala
  - IDRC-Infectious Disease Research Collaboration, IDRC Tororo Hospital Station Road, Tororo

IPD SHARING:
Plan to Share IPD: Yes
All IPD data that underlie the results presented herein
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of the study completion date
Access Criteria: Anonymized participant-level data may be shared with external researchers in accordance with trial participants' written and executed informed consent and applicable local regulations. Qualified researchers may submit a request along with a research proposal to Gates MRI for review. A data sharing agreement must be in place before any clinical trial data are shared. Additional restrictions may apply due to contractual obligations or regulatory constraints.